CLINICAL TRIAL: NCT00011102
Title: Prevention of Weight Gain in Women Aged 25 Through 44
Brief Title: Prevention of Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: Klem (completed); DK53942
Record Dates: First submitted 2001-02-09; First posted 2001-02-09 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Body Weight Changes
Keywords: weight gain
MeSH Terms: conditions — Obesity; Body Weight Changes; Weight Gain

INTERVENTIONS:
Behavioral: Weight Gain Prevention for Women Project

SUMMARY:
The purpose of this study is to test methods for preventing weight gain in normal-weight and overweight women aged 25 through 44. Participants will complete brief questionnaires about their health, eating and exercise habits, and use of weight control strategies. They will then be randomly assigned to 1 of 3 treatment conditions. All 3 treatments receive information on the importance of maintaining a healthy body weight, the components of a healthy diet, and ways to increase activity levels. The 3 treatment differ in how this information is delivered. At 12, 24 and 36 months after enrolling in the study, participants will attend assessment sessions. They will complete questionnaires and have body weight measured.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 21 through 30

Exclusion Criteria:

* Presence of chronic disease that precludes regular physical activity or changes in dietary intake
* Currently receiving treatment for psychological disorder
* Currently pregnant or having given birth within last 12 months
* Use in last 3 months of weight loss medications or other drugs that affect body weight
* Participation in a weight loss program in last 12 months
* Planning to relocate outside the study area in the next 3 years

Ages: 25 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2001-02; Study Completion 2001-12

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States